CLINICAL TRIAL: NCT03107455
Title: European Registry of MitraClip in Acute Myocardial Infarction
Brief Title: MitraClip in Acute Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: Fundación Investigación Sanitaria en León (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Felipe Fernandez Vazquez, MD PhD, Fundación Investigación Sanitaria en León
Other Study IDs: EREMMI
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Mitral Regurgitation; Acute Myocardial Infarction
Keywords: MitraClip; Acute mitral regurgitation; Acute myocardial infarction
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: MitraClip — MitraClip consists in two clip arms and opposing grippers, which can be opened and closed against each other in order to grasp and gain cooptation of MV leaflets at the origin of the regurgitant jet

SUMMARY:
Acute MR may develop in the setting of an acute myocardial infarction (AMI) as a result of papillary muscle dysfunction or rupture, and these patients are grossly underrepresented in MitraClip registries. Our group has recently published the Spanish experience with MitraClip in acute MI, but only 5 patients could be collected. However, the results of our initial experience are highly encouraging since patients performed well in such life-threatening condition. In order to expand the information of the device in this condition, our aim is to start a multinational registry in Europe.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 year-old
* Transmural myocardial infarction in the previous 4 weeks (managed under current guideline's recommendations).
* Symptomatic severe mitral regurgitation diagnosed by left ventriculography, transthoracic echo or trans-oesophageal echo. Symptoms may vary form heart failure to cardiogenic shock.
* Symptoms should be stabilized by medical management: iv diuretics, inotropic support, LV assistance devices
* Considered by heart team at high risk for conventional surgery

Exclusion Criteria:

* Anatomy not suitable for MitraClip implantation
* Technical contraindication for access to left atrium
* Patient candidate for emergent heart transplant
* Uncontrolled infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing transmural myocardial infarction in the previous 4 weeks and developing secondary mitral regurgitation not responding to medical therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Composite primary end point | 6 month
  death from cardiac causes, readmission due to heart failure and mitral regurgitation >2+

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Estevez-Loureiro, PhD, Principal Investigator — University Hospital Leon; Carmelo Grasso, PhD, Principal Investigator — Ferraroto Hospital Catania; Jan Van der Heijden, PhD, Principal Investigator — St. Antonius Hospital

IPD SHARING:
Plan to Share IPD: No